CLINICAL TRIAL: NCT04290702
Title: The Effect of Epidural, Combined and Dural Puncture Labor Epidural on Pain, Analgesics and Course of Vaginal Delivery: Randomised, Double Blind Study
Brief Title: Comparison of Epidural, Combined and Dural Puncture Labor Epidural on Pain, and Course of Vaginal Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Staikou Chryssoula, Associate Professor, University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 155/19-12-19
Record Dates: First submitted 2020-01-19; First posted 2020-03-02 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Labor Pain; Analgesia
MeSH Terms: conditions — Labor Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: 3 groups with different regional analgesic technique
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- epidural (Active Comparator)
  Interventions: Procedure: regional analgesia for labor
- combined (Active Comparator)
  Interventions: Procedure: regional analgesia for labor
- dural puncture epidural (Active Comparator)
  Interventions: Procedure: regional analgesia for labor

INTERVENTIONS:
Procedure: regional analgesia for labor — three commonly used regional analgesic techniques are used, with local anesthetic ropivacaine, opioid fentanyl, parturient controlled epidural analgesia

SUMMARY:
The three standard techniques used for labor analgesia, thus epidural, combined spinal-epidural and dural puncture epidural will be compared regarding their impact on pain intensity, analgesic and local anesthetic consumption and course of vaginal delivery in a prospective, randomised, double blind manner

ELIGIBILITY:
Inclusion Criteria:

* parturients requiring regional labor analgesia
* dilation less than 5cm

Exclusion Criteria:

* contraindication for regional technique
* refuse to participate
* language barriers
* obesity
* no pain

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
analgesic consumption | during the procedure/delivery
  the amount of local anesthetic and opioid that required during labor

SECONDARY OUTCOMES:
pain intensity on a numerical rating scale (minimum=0, maximum=10) | during the procedure/delivery
  pain intensity
duration of labor | until delivery
  duration of first stage
satisfaction on a numerical rating scale (minimum=0, maximum=10) | during the procedure/delivery
  satisfaction of parturients

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Aretaieio Hospital, University of Athens, Athens, Attica
  - Aretaieio Hospital, Athens